CLINICAL TRIAL: NCT01755728
Title: Paracetamol (Acetaminophen) for Closure of PDA in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Senior neonatologist, Hillel Yaffe Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 77-12-HYMC-CTIL
Record Dates: First submitted 2012-12-16; First posted 2012-12-24 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: PDA
Keywords: Paracetamol; Acetaminophen; PDA; Preterm infants
MeSH Terms: interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- No known PDA (No Intervention): For all infants, we do echo cardiogram study only if they are suspected of having PDA, due to sings and symptoms. Hence, we do not do echo cardiogram study to most of the infants.
- Ibuprofen (Active Comparator): If there is a PDA, that should be treated, and the infant is less than 2 weeks of age, we use ibuprofen, as this is the gold standard in literature.
  Interventions: Drug: Ibuprofen
- Surgical closure of PDA (Active Comparator): Infants with symptomatic PDA, who had to be treated, but could not be treated by ibuprofen, either due to age (> 2 weeks) or due ibuprofen contraindications (thrombocytopenia or renal failure), whose could not be treated by paracetamol (either because of parents' refuse or because they were on nothing per os protocol due to other disease), for whom surgery was the treatment of choice to close the arterial duct.
  Interventions: Procedure: Closure of PDA
- Paracetamol (Experimental): Infants with symptomatic PDA who could not be treated with ibuprofen, and their parents agreed and they could be treated with paracetamol.
  Interventions: Drug: Paracetamol
- DA closed spontaneously (No Intervention): Infants with PDA, who did not get any treatment for it, and the duct was closed spontaneously.

INTERVENTIONS:
Drug: Paracetamol — Per gavage paracetamol 15 mg/kg every 6 hours, for up to 7 days.
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Ibuprofen — Per Gavage ibuprofen 10mg/kg x 3/d for up to 5 days Gold standard per literature
  Arms: Ibuprofen
Procedure: Closure of PDA — Open surgery for closure of PDA
  Arms: Surgical closure of PDA

SUMMARY:
There is a report that acetaminophen may have a role in pharmacological closure of PDA (Patent arterial duct) in preterm infants.

The investigators conducted this open label non randomized and non control study to try to support that report.

DETAILED DESCRIPTION:
In-uteri, the arterial duct connects between the aorta and the main pulmonary artery, thus bypassing the lungs. Since the high pulmonary pressure and the low systemic pressure, the shunt trough the arterial duct in that time is right to left.

After birth, systemic pressure rises and pulmonary pressure declines. As oxygen saturation rises, and prostaglandin secretion, the arterial duct closes, usually. In preterm infants, the arterial duct may remain open after birth. At this tume the shunt would be left to right, that would cause pulmonary congestion, and systemic hypoperfusion.

Ibuprofen is the treatment of choice for PDA in preterm infants. Yet, ibuprofen is not effective after two weeks of age. Moreover, there are situations that prevent treatment with ibuprofen, such as thrombocytopenia or renal failure. Surgical closure of arterial duct is an alternative treatment, if ibuprofen is contraindicated, or if it fails.

Lastly, there was a report that acetaminophen may have a role in pharmacological closure of PDA in preterm infants.

The investigators conducted this open label non randomized and non control study to try to support that report.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with symptomatic PDA who could not be treated with ibuprofen

Exclusion Criteria:

* None

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Closure of arterial duct - yes / No | 1 week
  Echo-cardiogram that will give exact answer to the question: "was the arterial duct closed"?

SECONDARY OUTCOMES:
Need for surgical closure of arterial duct | 1 week
  The clinical state of the infant will guide the team to ask the parents and the chest surgeon to surgically close the arterial duct

OTHER OUTCOMES:
Death or deterioration | 1 week
  The infant state deteriorates so quickly that it will die, either because of complication of the arterial duct, or because other causes, such as sepsis, metabolic disorder, etc...

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe medical center, Hadera, Israel
Locations (1):
- Neonatal intensive care unit, Hillel Yaffe medical center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammerman C, Bin-Nun A, Markovitch E, Schimmel MS, Kaplan M, Fink D. Ductal closure with paracetamol: a surprising new approach to patent ductus arteriosus treatment. Pediatrics. 2011 Dec;128(6):e1618-21. doi: 10.1542/peds.2011-0359. Epub 2011 Nov 7. PMID 22065264
- [Background] Hammerman C, Bin-Nun A, Kaplan M. Managing the patent ductus arteriosus in the premature neonate: a new look at what we thought we knew. Semin Perinatol. 2012 Apr;36(2):130-8. doi: 10.1053/j.semperi.2011.09.023. PMID 22414884
- [Background] Oncel MY, Yurttutan S, Uras N, Altug N, Ozdemir R, Ekmen S, Erdeve O, Dilmen U. An alternative drug (paracetamol) in the management of patent ductus arteriosus in ibuprofen-resistant or contraindicated preterm infants. Arch Dis Child Fetal Neonatal Ed. 2013 Jan;98(1):F94. doi: 10.1136/archdischild-2012-302044. Epub 2012 May 18. No abstract available. PMID 22611117
- [Background] Peterson RG. Consequences associated with nonnarcotic analgesics in the fetus and newborn. Fed Proc. 1985 Apr;44(7):2309-13. PMID 3884385
- [Background] Rudolph AM. Effects of aspirin and acetaminophen in pregnancy and in the newborn. Arch Intern Med. 1981 Feb 23;141(3 Spec No):358-63. doi: 10.1001/archinte.141.3.358. PMID 7469626
- [Background] Simbi KA, Secchieri S, Rinaldo M, Demi M, Zanardo V. In utero ductal closure following near-term maternal self-medication with nimesulide and acetaminophen. J Obstet Gynaecol. 2002 Jul;22(4):440-1. doi: 10.1080/01443610220141489. No abstract available. PMID 12521476
- [Background] Weintraub A, Mankuta D. Dipyrone-induced oligohydramnios and ductus arteriosus restriction. Isr Med Assoc J. 2006 Oct;8(10):722-3. No abstract available. PMID 17125127
- [Background] Burdan F, Staroslawska E, Szumilo J. Prenatal tolerability of acetaminophen and other over-the-counter non-selective cyclooxygenase inhibitors. Pharmacol Rep. 2012;64(3):521-7. doi: 10.1016/s1734-1140(12)70847-2. PMID 22814005